CLINICAL TRIAL: NCT04805138
Title: Influence of Soft Tissue Thickness Upon Dental Implant Esthetics
Status: Completed | Type: Observational
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Gonzalo Blasi, Clinical Instructor, Universitat Internacional de Catalunya
Other Study IDs: PER-ECL-2018-07
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Peri-implant Mucositis; Implant Complication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Spectrophotometer — To objectively measure the discoloration of the peri-implant mucosa, spectrophotometric measurements of the buccal mucosa will be performed at study implant and at control tooth.

SUMMARY:
Since the beginning of the implant dentistry, a large variety of materials have been used for restoring single or multiple implants, such as gold, titanium, alumina (Al2O3), and zirconia (ZrO2). Patient physical and esthetic requirements play one of the most important role in making decisions related to which material should be chosen. In fact, long-term stability, compatibility with oral tissues esthetics and costs should be considered. Several studies demonstrated that both titanium and zirconia have an excellent biocompatibility and long-term stability even though something could change in terms of esthetic outcomes. Related to esthetics, the color of the peri-implant mucosa is an essential factor that clinicians have to take in to account. Unfortunately, discoloration of peri-implant mucosa sometimes happens. Some authors hypothesized that titanium abutments could provoke a grayish appearance of the mucosa, and, in order to avoid this problem, other authors suggested to perform augmentation of the peri-implant soft tissue thickness in the esthetic area. A study on pig maxillae found that the type of abutment or crown material and the mucosa thickness have significant influences on color changes of the mucosa. Titanium induced the most prominent color change, and, in patients with thinner mucosa, zirconia induced the least noticeable color changes. Nowadays, to reliably evaluate differences in color in implantology, the most used method is spectrophotometry, due to the capacity of detecting even small color differences and due to the higher reproducibility. Several investigations on pig jaws using spectrophotometric measurements were carried out recently, with the aim of investigating the color changes. It was found that generally titanium abutment lead to a more pronounced discoloration; however, gingival thickness greater than 2 mm did not reveal any difference related to the type of abutments. In addition, an increase in mucosal thickness might minimize the discoloration. The only study on human patients revealed that the color of the peri-implant mucosa presents more dark, green and blue components compared to the natural gingiva. Soft tissue thickness appeared a crucial factor with respect to the spectrophotometrically measured degree of peri-implant mucosal discoloration, with a trend for less pronounced discolorations in patients with thick mucosa. Furthermore, the authors found that peri-implant mucosa was on average 0,5-0,7 mm thicker than natural gingiva. However, this study evaluated the thickness of the gingiva by means of CBCT, which could lead to some errors due to the superimposition of the lips and cheeks, as well as the tongue that occupies the most space of the oral cavity. Moreover, esthetics were evaluated by clinicians visually at a specific distance asking them if discoloration was visible or not visible. Furthermore, no questionnaire was given to patients to evaluate esthetics neither discomfort while brushing. Therefore, The objective of this cross-sectional study is to evaluate the influence of gingival thickness (GT) upon mucosal color (MC) around dental implants measured spectrophotometrically. A secondary goal is to evaluate the correlation between mucosal color changes and type of abutment material around dental implants.

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than18 years old,
* periodontally and systemically healthy
* presence of at least one dental implant placed on the upper anterior maxilla, with a follow-up period of at least 1 year after prosthesis delivery
* full-mouth plaque and bleeding score ≤20%; presence of adjacent teeth
* no signs of peri-implant inflammation
* bleeding on probing or suppuration
* complete medical and dental history report.

Exclusion Criteria:

* Lack or minimal keratinized mucosa (<2mm)
* patients with uncontrolled periodontal disease
* active orthodontic therapy
* restorations on contralateral teeth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with at least one dental implant in the anterior upper maxilla (right first premolar to left first premolar). They will be selected, on a consecutive basis, among individuals referred to the periodontology department clinic floor.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
The influence of gingival thickness (GT) upon mucosal color (MC) around dental implants measured spectrophotometrically | At least 1 year after definitive crown in place.

SECONDARY OUTCOMES:
A secondary goal is to evaluate the correlation between mucosal color changes and type of abutment material around dental implants. | At least 1 year after definitive crown in place.

CONTACTS AND LOCATIONS:
Locations (1):
- International University of Catalunya, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided